

## **UNIVERSITY OF OXFORD**



Neurosciences Building Department of Psychiatry Warneford Hospital Oxford, OX3 7JX

Tel. (01865) 618324 Fax. (01865) 251076

E-mail: amy.gillespie@psych.ox.ac.uk

## **INFORMED CONSENT FORM (ICF)**

Title of Project: The effect of PF-04995274 on emotional processing in un-medicated depressed patients

Please Initial Box if you agree

| 1. I confirm that I have read and understand the participant information sheet dated 21/02/2017 (version 1.5) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. |
|---|
| 2. I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. |
| 3. I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from University of Oxford, from regulatory authorities [and from the NHS Trust(s)], where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. |
| 4. I give permission for my general practitioner to be contacted regarding my participation in the study. |
| 5. I agree to donate (blood and urine samples). I consider these samples a gift to the University of Oxford and I understand I will not gain any direct personal or financial benefit from them. |
| 6. I understand that the information collected about me may be used in an anonymous form to support other research in the future. It will not be possible for me to be identified by it. |
| 7. I understand that this is a research scan that is not useful for medical diagnosis, and that scans are not routinely looked at by a doctor. If a concern is raised about a possible abnormality on my scan, I will only be informed if a doctor thinks it is medically important such that the finding has clear implications for my current or future health. |
| 8. I agree to take part in the above study. |

The effects of PF-04995274 on emotional processing in un-medicated depressed patients

Informed Consent Form (ICF), Version 1.2; 21/02/18

IRAS project ID: 237793

REC reference: 18/SC/0076 Page 1 of 2

| Additional: | | | |
|---|---|---|---|
| I agree to be contacted about ethically approved research studies for which I may be suitable. | | Yes | No |
| I understand that agreeing to be co<br>studies. | ontacted does not oblige me | to participate in any further | |
| Name of Participant | Signature | Date | |
| Name of person taking consent | Signature | <br>Date | |

REC reference: 18/SC/0076 Page 2 of 2